CLINICAL TRIAL: NCT02536040
Title: Pragmatic Trial of Topical Diammine Silver Fluoride for Dental Caries Arrest
Brief Title: Stopping Cavities Study: Diammine Silver Fluoride
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advantage Dental Services, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 003
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Results first posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2016-08

CONDITIONS: Dental Caries
Keywords: silver diamine fluoride; diammine silver fluoride; children
MeSH Terms: conditions — Dental Caries | interventions — silver fluoride; silver diamine fluoride; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 38% diamine silver fluoride (Experimental): Topical application of 38% diammine silver fluoride to active cavity
  Interventions: Drug: 38% diammine silver fluoride
- Water (Placebo Comparator): Topical application of fluoride free water to active cavity
  Interventions: Other: Water

INTERVENTIONS:
Drug: 38% diammine silver fluoride — treatment of cavity with study agent
  Other Names: silver fluoride; silver diamine fluoride
  Arms: 38% diamine silver fluoride
Other: Water — Fluoride free, distilled water
  Arms: Water

SUMMARY:
This study is being conducted to test whether the use of diammine silver fluoride (also called silver diamine fluoride) hardens the cavity sufficiently so that it arrests.

DETAILED DESCRIPTION:
Phase III RCT with two arms: (1) 38% diammine silver fluoride; (2) distilled fluoride free water. Subjects are 200 preschool children in good general health with untreated tooth decay. Intervention is topical application of the study drug to the open cavity. Primary outcome is caries activity at 14-21 days.

ELIGIBILITY:
Inclusion Criteria:

* Nyvad criteria 3
* Active carious lesion

Exclusion Criteria:

* Allergy to silver
* Stomatitis or oral ulcerative condition
* Weight less than 15 kg

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milgrom, DDS, Study Director — Advantage Dental Plans
Locations (1):
- Advantage Dental Plans, Redmond, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 38% Diamine Silver Fluoride | Water
Started | 30 | 36
Completed | 29 | 35
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 38% Diamine Silver Fluoride | Water | Total
Number analyzed (Participants) | 30 | 36 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.7 (.6) | 4.9 (.5) | 4.8 (.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant without follow-up excluded from placebo group: male One participant without follow-up excluded: female
  Participants
    number analyzed (Participants) | 29 | 35 | 64
    Female | 13 | 18 | 31
    Male | 16 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant without follow-up excluded from placebo group: not hispanic or latino One participant without follow-up excluded from test group: hispanic or latino
  Participants
    number analyzed (Participants) | 29 | 35 | 64
    Hispanic or Latino | 15 | 23 | 38
    Not Hispanic or Latino | 14 | 12 | 26
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant without follow-up excluded from placebo: White One participant without follow-up excluded from test: White
  Participants
    number analyzed (Participants) | 29 | 35 | 64
    American Indian or Alaska Native | 2 | 0 | 2
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 27 | 33 | 60
    More than one race | 0 | 2 | 2
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: Two subjects excluded without follow-up: United States
  participants
    United States: number analyzed (Participants) | 29 | 35 | 64
    United States | 29 | 35 | 64

OUTCOME MEASURES:

1. Primary Outcome: Dental Caries Activity
Description: Proportion of treated teeth with active decay that were arrested by the treatment measured using the Nyvad criterion code 6 reflecting hardness of the lesion and color change
Time Frame: 14-21 days
Measure: Mean (Standard Deviation); unit: Proportion of arrested caries lesions
Arm/Group | 38% Diamine Silver Fluoride | Water
Number analyzed (Participants) | 29 | 35
Proportion of arrested caries lesions | .72 (.38) | .05 (.18)

ADVERSE EVENTS:
Time Frame: The primary focus of the adverse events clinical examination was to detect intramural soft tissue changes 2 days following the localized treatment of the teeth. It was not measured 14-21 days later when the primary outcome was assessed.
Description: Primary focus of adverse event assessment was intramural changes associated with the localized topical treatment of the teeth ((infection, inflammation, ulceration).
Arm/Group | 38% Diamine Silver Fluoride | Water
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/35
Other Adverse Events (participants affected / at risk) | 0/29 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No